CLINICAL TRIAL: NCT07383337
Title: A Randomized, Double-blind Crossover Pilot Trial to Compare the Olfactory Perception of a Fragrance-Loaded SpECs Over Time
Brief Title: Comparing the Olfactory Perception of a Fragrance-Loaded SpECs Over Time
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons in Ireland - Medical University of Bahrain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 271/20-May-2025
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Perception, Self
Keywords: fragrance; SpECs; Olfactory
MeSH Terms: conditions — Anosmia | interventions — Odorants

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Pilot randomized, double-blind crossover trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Fragrance loaded with a concentration of SpECs grains. (Experimental): Fragrance delivery system: SpECs loaded with fragrance (50mg/ml perfume)
  Interventions: Other: Fragrance
- Group B: Fragrance loaded without SpECs grains (Active Comparator): fragrance without SpECs
  Interventions: Other: Fragrance

INTERVENTIONS:
Other: Fragrance — this intervention involves the controlled use of specific fragrance with and withouth SpECs grains

SUMMARY:
The human olfactory system plays a crucial role in sensory perception, influencing emotional states, memory, and interpersonal interactions(1). Fragrance durability and intensity are critical factors in the evaluation of perfumes and other scented products. The ability of fragrance formulations to maintain consistent scent intensity over time is a major contributor to a product's overall efficacy and consumer satisfaction,

Primary Aim To compare the perceived strength of a topical fragrance delivered via SpECs across a period of 8 hours using subjective ratings by participants and an independent examiner.

Objectives

1. To investigate whether the encapsulated fragrance intensity, as perceived by participants, decreases less over time compared with fragrance alone, after application to the skin.
2. To investigate whether the encapsulated fragrance intensity, as perceived by an independent examiner, decreases less over time compared with fragrance alone, after application to the skin.

DETAILED DESCRIPTION:
The human olfactory system plays a crucial role in sensory perception, influencing emotional states, memory, and interpersonal interactions(1). Fragrance durability and intensity are critical factors in the evaluation of perfumes and other scented products. The ability of fragrance formulations to maintain consistent scent intensity over time is a major contributor to a product's overall efficacy and consumer satisfaction.

SporoSpECsin exine capsules (SpECs), are extracted from either pollen or plant spores in the form of empty porous microcapsules penetrated by nano-diameter sized channels. These channels enable a variety of active ingredients to be loaded into the SpECs chambers; hence, giving universality to the system to encapsulate such as a variety of antibody fragments, oils and proteins and peptides. The preparation that is to be used in this study has been provided to us as a gift by Sporomex Ltd, UK that is presently being used as a cosmetic preparation commercially, and has been investigated as a taste masking agent(2) and for oral pharmaceutical delivery(3).

It is unknown if fragrance loading of these SpECs will enhance the longevity of the fragrance on the skin. This study aims to evaluate the olfactory perception of a SpECs-based fragrance delivery system over an 8-hour period. The study will compare subjective ratings of the fragrance's intensity by participants and an independent examiner. This randomized, double-blind crossover trial will provide insights into the effectiveness of SpECs as a fragrance delivery medium, while also considering the influence of skin chemistry and time on olfactory perception. By eliminating patient variability, crossover studies can be more efficient than equivalently sized parallel group trials, where each participant receives only one treatment. Hence, treatment effects can be measured with greater accuracy using the same number of participants.

Type of Study Pilot randomized, double-blind crossover trial Participants

* Sample size: 10 female participants.
* Inclusion criteria:

  * Females aged between 18 and 45 years.
  * No history of olfactory impairment, allergies to pollen or fragrances, or skin conditions.
* Exclusion criteria:

  * Current use of medications that affect olfactory function (e.g., antihistamines).
  * Pregnancy or breastfeeding.
  * Any active upper respiratory tract infection within 2 weeks of the clinical trial
  * Any known skin allergy. Intervention
* Fragrance delivery system: SpECs loaded with fragrance (50mg/ml perfume) versus fragrance without SpECs
* Application: A smear layer of the fragrance-loaded SpECs will be applied to the wrist of each participant.

Randomization and Blinding

* Participants will be randomized into two groups:

  1. Group A: Fragrance loaded with a concentration of SpECs grains.
  2. Group B: Fragrance loaded without SpECs grains.
* Double-blinding: Neither the participants nor the independent examiner will know which preparation of the fragrance will be applied to the skin.

ELIGIBILITY:
Inclusion Criteria:

* Females aged between 18 and 45 years.
* No history of olfactory impairment, allergies to pollen or fragrances, or skin conditions.

Exclusion Criteria:

* Current use of medications that affect olfactory function (e.g., antihistamines).
* Pregnancy or breastfeeding.
* Any active upper respiratory tract infection within 2 weeks of the clinical trial
* Any known skin allergy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participation is limited to females, as the intervention focuses on factors specifically related to women's perception of fragrance.
Enrollment: 10 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Sustained olfactory perception over time. | 6 hour period- 4 timepoints
  The study will determine whether fragrance-loaded SpECs provides a sustained olfactory perception over time.

SECONDARY OUTCOMES:
Impact of SpECs concentration on fragrance | 6 hour period- 4 timepoints
  Insights into the impact of SpECs concentration on fragrance strength and duration will be obtained.
alignment between participant's and independent examiner's ratings | 6 hour period- 4 timepoints
  The alignment between participant's subjective ratings and the independent examiner's ratings will help validate the reliability of self-assessments in olfactory studies.

CONTACTS AND LOCATIONS:
Overall Officials: Mariam Murad, Principal Investigator — Royal College of Surgeons, Ireland

REFERENCES:
- [Background] Herz RS. The Role of Odor-Evoked Memory in Psychological and Physiological Health. Brain Sci. 2016 Jul 19;6(3):22. doi: 10.3390/brainsci6030022. PMID 27447673
- [Background] Diego-Taboada A , Maillet L , Banoub JH , Lorch M , Rigby AS , Boa AN , Atkin SL , Mackenzie G . Protein free microcapsules obtained from plant spores as a model for drug delivery: ibuprofen encapsulation, release and taste masking. J Mater Chem B. 2013 Feb 7;1(5):707-713. doi: 10.1039/c2tb00228k. Epub 2012 Nov 27. PMID 32260776
- [Background] Wakil A, Mackenzie G, Diego-Taboada A, Bell JG, Atkin SL. Enhanced bioavailability of eicosapentaenoic acid from fish oil after encapsulation within plant spore exines as microcapsules. Lipids. 2010 Jul;45(7):645-9. doi: 10.1007/s11745-010-3427-y. Epub 2010 May 22. PMID 20495964